CLINICAL TRIAL: NCT04870541
Title: Comparative Study Between Nefopam and Ondansteron for Prevention of Post Spinal Shivering. A Randomized Controlled Trial.
Brief Title: Nefopam Versus Ondansteron for Prevention of Post Spinal Shivering.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HDF15891
Record Dates: First submitted 2021-03-30; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Shivering; Adverse Effects in the Therapeutic Use of Anaesthetic
MeSH Terms: interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients receiving Ondansetron (Active Comparator)
  Interventions: Drug: Ondansetron 8mg
- Patients receiving Nefopam (Active Comparator)
  Interventions: Drug: Nefopam Injectable Solution

INTERVENTIONS:
Drug: Ondansetron 8mg — Patients receiving 8 mg of ondansetron diluted in 20 ml of 0.9% normal saline over 30 minutes as they arrive to the operating theater(75 patients).
  Arms: Patients receiving Ondansetron
Drug: Nefopam Injectable Solution — Patients receiving 20 mg of nefopam diluted in 20 ml of 0.9% normal saline over 30 minutes as they arrive to the operating theater (75 patients)
  Arms: Patients receiving Nefopam

SUMMARY:
Spinal anesthesia affects the homeostatic systems resulting in intraoperative hypothermia and subsequently shivering. In fact, shivering may be seen after this technique in 30 to 40% of cases . Ondansetron and Nefopam have been used to prevent intraoperative shivering . However, no prospective, randomized, double-blind study has been conducted to this date in order to compare nefopam with ondansetron in the prevention of post-spinal anesthesia shivering.

The primary objective of this prospective, randomized, double-blind study is to compare the incidence and intensity of shivering after spinal anesthesia for non-obstetric surgery in 2 groups of patients.

Group A: Patients receiving 8 mg of ondansetron diluted in 20 ml of 0.9% normal saline over 30 minutes as they arrive to the operating theater(75 patients).

• Group B: Patients receiving 20 mg of nefopam diluted in 20 ml of 0.9% normal saline over 30 minutes as they arrive to the operating theater (75 patients)

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* scheduled for a surgery under spinal anesthesia

Exclusion Criteria:

* pregnant or breastfeeding (for the women), if they are
* Allergy to any of the drugs to be used
* Long QT syndrome
* Hepatic insufficiency
* Renal failure
* Parkinson's disease
* Epilepsy
* Glaucoma
* Phenylketonuria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of shivering | Shivering score was noted every 15 minutes from drug administration up to 120 minutes.
  Number of episodes of shivering and variation will be noted every 15 minutes from drug administration up to 120 minutes.
Grade of shivering | Shivering score was noted every 15 minutes from drug administration up to 120 minutes.
  Grades of shivering will be noted every 15 minutes from drug administration up to 120 minutes. Shivering will be graded : 0 = no shivering, 1= piloerection or peripheral vasoconstriction but no visible shivering, 2 = muscular activity in only one muscle group, 3 = muscular activity in more than one muscle group but not generalized shivering, 4 = shivering involving the whole body.

SECONDARY OUTCOMES:
Nausea/Vomitting | Every 15 minutes from drug administration up to 120 minutes
  Number of episodes of nausea and/or vomiting during and after surgery.
Hypotention/Bradycardia | Every three minutes from drug administration up to 120 minutes.
  Hypotention: Number of episodes of hypotension SBP <90mmhg or <25% of baseline SBP in post spinal anesthesia until discharge from the PACU.
  Bradycardia: Number of episodes of bradycardia <50 / min post-spinal anesthesia until discharge from the PACU.
Pain on injection site by analogue visual scale. | During administration of drug.
  Pain upon administration of drug on site of injection will be assessed using the analogue visual scale .

CONTACTS AND LOCATIONS:
Locations (1):
- Universite Saint Joseph , Hotel Dieu de France, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang P, Park SK, Yoo S, Hur M, Kim WH, Kim JT, Bahk JH. Comparative effectiveness of pharmacologic interventions to prevent shivering after surgery: a network meta-analysis. Minerva Anestesiol. 2019 Jan;85(1):60-70. doi: 10.23736/S0375-9393.18.12813-6. Epub 2018 Sep 18. PMID 30226340
- [Background] Crowley LJ, Buggy DJ. Shivering and neuraxial anesthesia. Reg Anesth Pain Med. 2008 May-Jun;33(3):241-52. doi: 10.1016/j.rapm.2007.11.006. PMID 18433676
- [Background] Mathews S, Al Mulla A, Varghese PK, Radim K, Mumtaz S. Postanaesthetic shivering--a new look at tramadol. Anaesthesia. 2002 Apr;57(4):394-8. doi: 10.1046/j.1365-2044.2002.2457_3.x. PMID 11949644
- [Background] Lv M, Wang X, Qu W, Liu M, Wang Y. Nefopam for the prevention of perioperative shivering: a meta-analysis of randomized controlled trials. BMC Anesthesiol. 2015 Jun 9;15:87. doi: 10.1186/s12871-015-0068-y. PMID 26055978
- [Background] Rai S, Verma S, Pandey HP, Yadav P, Patel A. Role of butorphanol and ondansetron premedication in reducing postoperative shivering after general and spinal anesthesia: A randomized comparative study from North India. Anesth Essays Res. 2016 May-Aug;10(2):319-23. doi: 10.4103/0259-1162.172724. PMID 27212768
- [Background] Marashi SM, Soltani-Omid S, Soltani Mohammadi S, Aghajani Y, Movafegh A. Comparing Two Different Doses of Intravenous Ondansetron With Placebo on Attenuation of Spinal-induced Hypotension and Shivering. Anesth Pain Med. 2014 Mar 18;4(2):e12055. doi: 10.5812/aapm.12055. eCollection 2014 May. PMID 24790900
- [Background] Tsai YC, Chu KS. A comparison of tramadol, amitriptyline, and meperidine for postepidural anesthetic shivering in parturients. Anesth Analg. 2001 Nov;93(5):1288-92. doi: 10.1097/00000539-200111000-00052. PMID 11682416